CLINICAL TRIAL: NCT02792530
Title: Daily Sodium Intake in Anuric Hemodialysis Patients and Interdialytic Weight Gain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0654-15-RMC
Record Dates: First submitted 2016-04-12; First posted 2016-06-07 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-04

CONDITIONS: End Stage Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- arm 1 (Other): Unuric hemodialytic patients who accumulate above 2.5 (4%) in intradialytic intervals before the nutritional intervention.
  Interventions: Other: Dietary consultation

INTERVENTIONS:
Other: Dietary consultation — Dietary consultation for sodium restriction to decrease dietary intake to 2 grams/day less than the patients consume currently

SUMMARY:
This study will evaluate the efficiency of dietary intervention on intradialytic weight gain. Uniric hemodialysis patients without serious dietary complications, who accumulate above 2.5 kg (or above 4%) of their dry weight, will undergo a series of dietary consultations for sodium restriction. One month after the intervention, their intradialytic weight accumulation will be measured.

DETAILED DESCRIPTION:
Inter Dialytic Weight Gain (IDWG) ascribed to fluid retention is one of the major clinical problem that patients in hemodialysis need to cope with between 2 subsequent hemodialysis especially in patients with no residual renal function. Fluid retention is associated with morbid conditions such as lower-extremity edema, ascites, pulmonary vascular congestion or edema, hypertension, and worsening heart failure. Gain weight above 2 kg between 2 subsequent hemodialysis found to be in higher risk of all-cause mortality and cardiovascular death .Lowering daily sodium intake found to mitigate fluid retention ,however there are only a few researches that check it. 2IDWG also associated with poorer quality of life. Dietary sodium restriction recommendation since the beginning of hemodialysis are based on association of this restriction with balance of hypertension and fluid retention. Sodium intake recommended for patients in hemodialysis is limited to 2 grams a day. Nevertheless, there are only a few studies that examine the efficiency of this restriction because of the complexity of measurement of sodium intake. One recently published study which used a 24-h recall to measure sodium intake, found a direct correlation between IDGW and mortality form any reason. In spite of this complexity, IDWG has been found to be in a direct relation with patients' nutrition status.

One of sodium-related issues is malnutrition. Malnutrition in dialysis is a risk factor for patients' morbidity and mortality. Higher sodium intake is associated with higher calorie and protein intake, while adherence to restriction of sodium intake is poor in hemodialysis. This is a reason for high importance to study effects of sodium restriction in people with more than 2.5 kg (or 4% of dry body weight) IDWG while following up their nutritional status

ELIGIBILITY:
Inclusion Criteria:

1. Adults >18 years providing signed informed consent.
2. Any patient more than 3 months in hemodialysis who reach his assigned dry weight.
3. Intradialytic weight gain of more than 2.5 liters or 4% of dry body weight in two mid-week sessions.
4. residual renal function of less than 200 ml per 24 hr.
5. expected to stay on hemodialysis for at least 6 month.

Exclusion Criteria:

1. Malnutrition as assessed by SGA: score C.
2. Dementia
3. Active malignancy
4. Active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Reduction in intradialytic weight gain (IDWG) | between baseline and 6 weeks
  Reduction in the weight gain at 2 subsequent hemodialysis in KG/

SECONDARY OUTCOMES:
dietary sodium intake. | at baseline and 6 weeks
  as measured by food recall assesment
Change in CRP values | between baseline and 6 weeks
Changes in subjective global assesment (SGA) | between baseline and 6 weeks
  SGA is a nutritional assesment measure
change in predialysis blood pressure | between baseline and 6 weeks
Changes in quality of life | between baseline and 6 weeks
  assessed by SF 36
number of hypotensive episode during dialysis | at baseline and 6 weeks
  define as drop of more than 20 mm hg systolic blood pressure from baseline